CLINICAL TRIAL: NCT01247233
Title: Phase III Multicentric Trial Comparing Accelerated Partial Breast Irradiation (APBI) Versus Standard or Hypofractionated Whole Breast Irradiation in Low Risk of Local Recurrence of Breast Cancer
Brief Title: Standard or Hypofractionated Radiotherapy Versus Accelerated Partial Breast Irradiation (APBI) for Breast Cancer
Acronym: SHARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTS02-SHARE; 2010-A00243-36 (Other: ID-RCB); UC-0140/1001 (Other: UNICANCER); RTS02 / SHARE (Other: UNICANCER)
Record Dates: First submitted 2010-10-26; First posted 2010-11-24 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Lumpectomy
Keywords: breast cancer; Accelerated Partial Breast Irradiation; invasive cancer; Hypofractionated Irradiation; Lumpectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard or Hypofractionated radiotherapy (Active Comparator): Whole breast RT, 50 Gy + "boost" 16 Gy. Whole breast hypofractionated RT without boost, either 40 Gy or 42.5 Gy
  Interventions: Radiation: Whole Breast Irradiation + Boost or Hypofractionated irradiation
- Accelerated Partial Breast Irradiation (APBI) (Experimental): APBI using 3D CRT technique, in 5 days, 38.5 Gy to the tumor bed
  Interventions: Radiation: Accelerated partial breast irradiation

INTERVENTIONS:
Radiation: Whole Breast Irradiation + Boost or Hypofractionated irradiation — Whole Breast Irradiation 50 Gy + Boost 16 Gy or Whole breast, either 40 Gy in 15 fractions in 3 weeks or 42.5 Gy in 16 fractions in 3 weeks
  Other Names: Standard radiation
  Arms: Standard or Hypofractionated radiotherapy
Radiation: Accelerated partial breast irradiation — Tumor bed 40 Gy in 10 fractions, 2 fractions of 4 Gy per day in 5 to 7 days.
  Other Names: APBI
  Arms: Accelerated Partial Breast Irradiation (APBI)

SUMMARY:
The standard treatment for localized breast cancer is based on conservative surgery (when possible) followed by radiation therapy (RT) delivered to the whole breast. The recommended total RT dose is 45 to 50 Gy delivered in 4.5 to 5 weeks followed by a 10 to 16 Gy boost to the tumor bed for 1 to 1.5 weeks. The rationale for the development of APBI was based on the difficulty for many patients to reach RT centers to receive standard whole breast irradiation (WBI) after conservative surgery. APBI offers decreased overall treatment time and several theoretical advantages over WBI, including a decrease in dose delivered to uninvolved portions of the breast and adjacent organs. If equivalence between the two treatments can be shown, then APBI will be considered as a historic evolution in breast cancer management.

In this phase III trial, designed in postmenopausal women >50 years of age, the objective is to compare the effectiveness and safety of APBI compared with whole breast irradiation. This study is also designed to ensure high quality criteria for surgery, pathology and RT techniques in the 3 arms and will allow to provide data on economics and costs.

DETAILED DESCRIPTION:
Following breast conservative surgery, patients will be stratified according to the following prognostic factors using a minimisation technique: age (<70 vs ≥70), HER2 status (HER2+ vs HER2-), hormonal receptor status (RH+ vs RH-) and lymph node invasion (pN0 vs pN0i+).

Patients will be allocated to receive either standard treatment, hypofractionated treatment or APBI.

Radiation therapy should be started between 4 and 12 weeks after the last surgery.

Patients treated with standard whole breast irradiation will receive a total dose of 50 Gy in 25 fractions, 2 Gy per day, 5 days a week. The boost of 16 Gy will be delivered in 8 fractions for all patients after completion of the 50 Gy, without interruption. All patients will receive one fraction per day, 5 fractions a week.

Patients treated with hypofractionated irradiation will receive a total dose of either 40 Gy (in 15 fractions, 2.66 Gy per day) or 42.5 Gy (in 16 fractions, 2.65 Gy per day) 5 days a week.

Patients treated with APBI will receive a total dose of 40 Gy in 10 fractions, delivered twice a day over a time period of 5-7 days. Each daily dose must be separated by 6 hours.

Patients will be followed at 3 and 6 month after the last dose of irradiation, at 12 months after the date of last surgery and then on a yearly basis during 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥50 years
* Menopausal status confirmed
* Pathology confirmation of invasive carcinoma (all types)
* Complete tumor removal and conservative surgery
* Pathologic tumor size of invasive carcinoma ≤2 cm (including the in situ component) pT1
* All histopathologic grades
* Clear lateral margins for the invasive and in situ disease (>2 mm)
* pN0 or pN(i+)
* No metastasis
* Radiotherapy should be started more than 4 weeks and less than 12 weeks after last surgery
* Surgical clips (4 to 5 clips in the tumor bed)
* No prior breast or mediastinal radiotherapy
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Information to the patient and signed informed consent

Exclusion Criteria:

* Multifocal invasive ductal carcinoma defined as the presence of at least two distinct tumors that are separated by normal tissue or when the distance between the two lesions does not permit conservative surgery
* Bilateral breast cancer
* No or less than 4 surgical clips in the tumor bed
* Nodal involvement : pN1 (including micrometastasis, mi+), pN2, pN3
* Metastatic disease
* internal mammary node involvement or supraclavicular lymph node involvement
* Indication of chemotherapy or trastuzumab
* Involved or close lateral margins for the invasive and /or in situ components (<2 mm) AND impossibility to re-operate or impossible to perform another conservative surgery
* Patients with known BRCA1 or BRCA2 mutations
* Previous mammoplasty
* Previous homolateral breast and/or mediastinal irradiation
* Previous invasive cancer (except basocellular epithelioma or in situ carcinoma of the cervix)
* No geographical, social or psychologic reasons that would prevent study follow

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Actual)
Dates: Start 2010-12-27 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
rate of local recurrence | 5 years
  To estimate and compare the rate of local recurrence between the experimental and control arms.

SECONDARY OUTCOMES:
Ipsilateral breast recurrence-free survival | 10 years
  To evaluate Ipsilateral breast recurrence-free survival
Nodal regional recurrence-free survival | 10 years
  To evaluate nodal regional recurrence-free survival
Distant recurrence-free survival | 10 years
  To evaluate distant recurrence-free survival
Disease-specific survival | 10 years
  To evaluate disease-specific survival
Overall survival | 10 years
  To evaluate the overall survival
Toxicities: Measurement of the rate and type of toxicity (acute and late toxic effects) | 10 years
  To evaluate rates and type of acute and late toxicities
Cosmetic: comparison of the cosmetic result (according to both the physician and the patient) | 10 years
  To evaluate Cosmetic results (Patient and Physician evaluations)
Quality of Life and Satisfaction | 10 years
  To evaluate the patient quality of life and patient satisfaction
Medico-economic study | 3 years
  To evaluate the cost of APBI compared with Standard and Hypofractionated irradiation

CONTACTS AND LOCATIONS:
Overall Officials: Yazid Belkacemi, MD PhD, Principal Investigator — Henri Mondor Hospital AP-HP, Créteil, France; Eric Lartigau, MD, Principal Investigator — Oscar Lambret Hospital, Lille, France; Céline Bourgier, MD, Principal Investigator — Institut de Cancérologie de Montpellier, Montpellier, France
Locations (34):
- France (34):
  - Centre de traitement des Hautes energie - Clinique de l'Europe, Amiens
  - Centre Hospitalier Universitaire, Amiens
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier, Brivé
  - Centre Francois Baclesse, Caen
  - CH Chambery, Chambéry
  - Hopital Henri Mondor, Créteil
  - Centre Leonard de Vinci, Dechy
  - CHU Michallon, Grenoble
  - Hôpital Robert Boulin, Libourne
  - Centre Oscar Lambret, Lille
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Clinique du Pont de Chaume, Montauban
  - Centre Hospitalier, Montélimar
  - CRLC Val d'Aurelle, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre d'Oncologie de Gentilly, Nancy
  - Clinique Hartmann, Neuilly-sur-Seine
  - Centre de Haute Energie, Nice
  - Groupe Hospitalier Pitié Salpétrière, Paris
  - Hopital Tenon, Paris
  - Saint Louis Hospital, Paris
  - Centre Catalan d'Oncologie, Perpignan
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - CH de Roanne, Roanne
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Paul Stauss, Strasbourg
  - Centre Marie Curie, Valence
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Derived] Belkacemi Y, Bourgier C, Kramar A, Auzac G, Dumas I, Lacornerie T, Mege JP, Mijonnet S, Lemonnier J, Lartigau E. SHARE: a French multicenter phase III trial comparing accelerated partial irradiation versus standard or hypofractionated whole breast irradiation in breast cancer patients at low risk of local recurrence. Clin Adv Hematol Oncol. 2013 Feb;11(2):76-83. PMID 23598908